CLINICAL TRIAL: NCT05086614
Title: The Efficacy and Safety of Thymosin-alpha 1 Used for Adjuvant Treatment After Radical Resection of High-risk Stage II and Stage III Colorectal Cancer
Brief Title: Thymosin-alpha 1 for Adjuvant Treatment After Radical Resection of High-risk Stage II and III Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TARCRC
Record Dates: First submitted 2021-09-23; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-03

CONDITIONS: Stage II Colorectal Cancer; Stage III Colorectal Cancer
Keywords: colorectal cancer; adjuvant treatment; thymosin-alpha 1; disease-free survival
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Thymalfasin

STUDY DESIGN:
Intervention Model Description: Patients with pathological high-risk stage II and stage III colorectal cancer after radical resection were randomly allocated to receive thymosin-alpha 1 or not in a 1:1 ratio.
Who Masked: Outcomes Assessor
Masking Description: There is no masking for participants or investigators. The outcomes assessors will be blind for the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thymosin (Experimental): Patients with pathological high-risk stage II and stage III colorectal cancer after radical resection.
  Interventions: Drug: Thymosin Alpha1
- Observe (No Intervention): Patients with pathological high-risk stage II and stage III colorectal cancer after radical resection.

INTERVENTIONS:
Drug: Thymosin Alpha1 — Receive thymosin-alpha 1 1.6mg with subcutaneous injection, twice a week, for 6 months after radical resection.
  Other Names: Thymalfasin
  Arms: Thymosin

SUMMARY:
For high-risk stage II and stage III colorectal cancer, even after radical resection and postoperative adjuvant chemo/radiotherapy, 30-40% of patients will still have recurrence and metastasis. Thymosin-alpha 1 is believed to improve immunity and may help promote tumor immunity to reduce the incidence of recurrence and metastasis. This study hopes to verify the effecacy and safety of thymosin-alpha 1 for adjuvant treatment of high-risk stage II and stage III colorectal cancer after radical resection.

DETAILED DESCRIPTION:
Patients with pathological high-risk stage II and stage III colorectal cancer after radical resection were randomly allocated to receive thymosin-alpha 1 twice a week for 6 months (experimental group) or not (control group) in a 1:1 ratio. At the same time, all patients will receive chemo/radiotherapy according to the Chinese Standards for Diagnosis and Treatment of Colorectal Cancer. The primary endpoint is 3-year DFS rate.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer receiving radical resection
* Pathologically diagnosed with high-risk stage II or stage III
* Eastern Cooperative Oncology Group performance status of 0-2
* Adequate hepatic, renal, and hematologic function

Exclusion Criteria:

* Had previously taken any immune-promoting drugs
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate | 3 years
  percentage of patients who have no recurrence or metastases or death at 3 years after surgery.

SECONDARY OUTCOMES:
3-year overall survival rate | 3 years
  percentage of patients who are alive at 3 years after surgery.
rate of adverse events related to thymosin-alpha 1 | 6 months
  percentage of patients with adverse events related to thymosin-alpha 1, including fever, allergies, skin rash, liver and kidney damage

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided